CLINICAL TRIAL: NCT02901080
Title: Naturalistic Study of Alpha-Stim in Patients With a Primary Working Diagnosis of Moderate-to-severe Generalised Anxiety Disorder Who Did Not Improve With Low Intensity Psychological Therapy Intervention
Brief Title: Clinical and Cost Effectiveness of Alpha-Stim AID CES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Electromedical Products International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206555
Record Dates: First submitted 2016-09-01; First posted 2016-09-15 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Pregnancy Tests; Patient Health Questionnaire; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cranial electrotherapy stimulation (Experimental): Alpha Stim AID cranial electrotherapy stimulation, Pregnancy test, Anxiety questionnaire, Quality of life questionnaire, Work and social questionnaire, Sleep questionnaire, Depression questionnaire, Quality of life and financial questionnaire
  Interventions: Device: Alpha Stim AID cranial electrotherapy stimulation; Behavioral: Pregnancy test; Other: Anxiety questionnaire; Other: Quality of life questionnaire; Other: Work and social questionnaire; Other: Sleep questionnaire; Other: Depression questionnaire; Other: Quality of life and financial questionnaire

INTERVENTIONS:
Device: Alpha Stim AID cranial electrotherapy stimulation — - 60 minutes of cranial electrotherapy stimulation via Alpha Stim AID once per day, for a minimum of 6 and maximum of 12 weeks.
Behavioral: Pregnancy test — - Pregnancy test x 1 (day 1)
Other: Anxiety questionnaire — - GAD-7 questionnaire x 6 (day 1, week 4, week 6, week 8, week 12 and week 24)
Other: Quality of life questionnaire — - EQ-5D-5L questionnaire x 6 (day 1, week 4, week 6, week 8, week 12 and week 24)
Other: Work and social questionnaire — - WASA questionnaire x 6 (day 1, week 4, week 6, week 8, week 12 and week 24)
Other: Sleep questionnaire — - Athens questionnaire x 6 (day 1, week 4, week 6, week 8, week 12 and week 24)
Other: Depression questionnaire — - PHQ-9 questionnaire x 6 (day 1, week 4, week 6, week 8, week 12 and week 24)
Other: Quality of life and financial questionnaire — - CSRI questionnaire x 3 (day 1, week 12 and week 24)

SUMMARY:
This is a single-centre research study in patients seen within an NHS Improving Access to Psychological Interventions (IAPT) service with suspected generalised anxiety disorder (GAD). The study will involve 120 patients from the Leicestershire and Rutland area in England, United Kingdom.

Participants will use the Alpha-Stim AID Cranial Electrotherapy Stimulations (CES) medical device, which is approved for use and proven to be safe and work for the treatment for anxiety, depression and insomnia.

Participants will use the Alpha-Stim AID for 60 minutes every day for 6 or 12 weeks, either whilst on the waiting list for standard care treatment from IAPT, or in conjunction with standard care treatment from IAPT.

The study will involve 6 study visits - one face-to-face at visit 1, followed by 5 visits via telephone at week 4, 6, 8, 12 and 24. At each visit, participants will be asked to complete questionnaires to assess anxiety, depression, sleep difficulty, quality of life and work and social functioning.

The purpose of the study is to gather evidence for the clinical benefits and cost effectiveness of the Alpha-Stim AID when used in an NHS setting - how well does it work, and does it's use result in cost savings for the NHS.

The study may show that the Alpha-Stim AID should be available on the NHS for patients with suspected GAD.

DETAILED DESCRIPTION:
Participants will have a baseline visit (day 1, visit 1) following identification as potentially eligible. The baseline visit will be face-to-face with a member of the research team, held at routine facilities used by the IAPT service. At the baseline visit, the participant will be consented for participation, have a urine pregnancy test first (if a female of child bearing potential) and the research team will administer the GAD-7 secondly, followed by EQ-5D-5L, WASA, PHQ-9, Athens, and CSRI surveys. Participants will then be instructed on how to use the Alpha-Stim AID device, and will have their first 60 minute, self-directed treatment session at home.

All further visits will be facilitated via telephone, scheduled between the research team and participant, within a 5 calendar day window of each time point.

At visit 2 (week 4), visit 3 (week 6), visit 4 (week 8), visit 5 (week 12) and visit 6 (week 24), the research team will administer the GAD-7, EQ-5D-5L, WASA, PHQ-9 and Athens. The CSRI will be repeated only at visit 5 and 6. Compliance with the 60 minute daily treatment session will also be assessed during the 6 or 12 week treatment window, in addition to any adverse events.

The 60-minute self-directed Alpha-Stim AID treatment sessions are undertaken at participant's home, on a daily basis for 6 weeks for all participants. During this 6-week period, participants will be on the waiting list for high intensity psychological therapy interventions.

Following 6 weeks of Alpha-Stim AID CES treatment, participants have the option to receive a further 6 weeks of treatment, which is likely to coincide with start of high intensity psychological therapy interventions as clinically indicated.

Following a maximum of 12 weeks' treatment with Alpha-Stim AID CES, all participants will cease to receive treatment on study.

All participants will continue to receive standard care assessment, as undertaken by the NHS IAPT service, standard care high intensity psychological therapy interventions as clinically indicated and provided by the NHS IAPT service, and standard care pharmacological treatments as prescribed by the participant's GP. Participation in this study will not influence nor compromise standard care treatment - all study procedures are additional to standard care. Participation in the study will have no impact upon the duration of the waiting time for high intensity psychological therapy interventions.

ELIGIBILITY:
Inclusion Criteria:

* Primary working diagnosis of moderate-to-severe GAD indicated via a GAD-7 score of 10 or more at baseline visit
* Previous treatment within an IAPT service with step two low intensity psychological therapy intervention
* Indicated for step three high intensity psychological therapy intervention and on the waiting list
* Capable of giving informed consent
* Female participants of child-bearing potential must have a negative urine human chorionic gonadotropin dipstick pregnancy test
* Female participants of child-bearing potential must be practising a highly effective method of contraception (failure rate of less than 1% per year when used consistently and correctly and agree to remain on a highly effective method throughout the 6 or 12 week treatment period. Examples of highly effective contraceptives include: barrier condoms, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), vasectomised partner, sexual abstinence (refraining from heterosexual intercourse), and oestrogen and progestogen containing hormonal contraception associated with ovulation.
* 18 years of age or above at baseline visit
* Able to understand written and verbal English

Exclusion Criteria:

* Primary working diagnosis of a mental disorder other than moderate-to-severe GAD (but other mental and anxiety disorders as secondary comorbidities is not an exclusion criteria)
* No previous treatment within an IAPT service with step two low intensity psychological therapy intervention
* Not indicated for step three high intensity psychological therapy intervention and not on the waiting list
* Requiring urgent clinical care
* Female participants of child-bearing potential with a positive urine human chorionic gonadotropin dipstick pregnancy test
* Female participants of child-bearing potential not willing to practice a highly effective method of contraception during the treatment period
* Implantation with a pace maker
* Implantation with an implantable cardioverter defibrillator (ICD)
* Incapable of giving informed consent
* 17 years of age or less at baseline visit
* Unable to understand written and verbal English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Morris, Professor, Principal Investigator — University of Nottingham
Locations (1):
- Leicestershire and Rutland Improving Access to Psychological Therapies (IAPT) Service, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data will form part of the final study report which will be used for submission to the UK National Institute for Clinical Excellence.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 161 participants who enrolled in the study began the treatment.
Groups:
- Cranial Electrotherapy Stimulation: Alpha Stim AID cranial electrotherapy stimulation, Pregnancy test, Anxiety questionnaire, Quality of life questionnaire, Work and social questionnaire, Sleep questionnaire, Depression questionnaire, Quality of life and financial questionnaire
  Alpha Stim AID cranial electrotherapy stimulation: - 60 minutes of cranial electrotherapy stimulation via Alpha Stim AID once per day, for 6 to 12 weeks.
  Pregnancy test: - Pregnancy test (day 1)
  Anxiety questionnaire: - GAD-7 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life questionnaire: - EQ-5D-5L (day 1, week 4, week 6, week 8, week 12 and week 24)
  Work and social questionnaire: - WASA (day 1, week 4, week 6, week 8, week 12 and week 24)
  Sleep questionnaire: - Athens (day 1, week 4, week 6, week 8, week 12 and week 24)
  Depression questionnaire: - PHQ-9 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life and financial questionnaire: - CSRI (day 1, week 12 and week 24)
Period: Overall Study
Arm/Group | Cranial Electrotherapy Stimulation
Started | 161
Completed | 112
Not Completed | 49

BASELINE CHARACTERISTICS:
Groups:
- Cranial Electrotherapy Stimulation: Alpha Stim AID cranial electrotherapy stimulation, Pregnancy test, Anxiety questionnaire, Quality of life questionnaire, Work and social questionnaire, Sleep questionnaire, Depression questionnaire, Quality of life and financial questionnaire
  Alpha Stim AID cranial electrotherapy stimulation: - 60 minutes of cranial electrotherapy stimulation via Alpha Stim AID once per day, for a minimum of 6 and maximum of 12 weeks.
  Pregnancy test: - Pregnancy test (day 1)
  Anxiety questionnaire: - GAD-7 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life questionnaire: - EQ-5D-5L (day 1, week 4, week 6, week 8, week 12 and week 24)
  Work and social questionnaire: - WASA (day 1, week 4, week 6, week 8, week 12 and week 24)
  Sleep questionnaire: - Athens (day 1, week 4, week 6, week 8, week 12 and week 24)
  Depression questionnaire: - PHQ-9 (day 1, week 4, week 6, week 8, wee
Arm/Group | Cranial Electrotherapy Stimulation
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.00 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 153
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 161

OUTCOME MEASURES:

1. Primary Outcome: Clinical Effectiveness in Generalised Anxiety Disorder Measured by at Least a 5 Point Reduction in Scores on the GAD-7
Description: The primary objective of this study is to evaluate the clinical effectiveness of treatment with Alpha-Stim AID Cranial Electrotherapy Stimulations (CES) for participants with a primary working diagnosis of generalised anxiety disorder (GAD), as defined by the NHS IAPT service in terms of reliable improvement (at least a 5 point improvement on the GAD-7),or recovery (total score of less than 7 and at least a 5 point improvement on the GAD-7), from baseline to week 24, following previous treatment with low intensity psychological therapy intervention.
Time Frame: 24 weeks
Population: Number of participants achieving at least 50% improvement on the GAD-7 from CES treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cranial Electrotherapy Stimulation at 100 uA for 60 Minutes: Alpha Stim AID cranial electrotherapy stimulation, Pregnancy test, Anxiety questionnaire, Quality of life questionnaire, Work and social questionnaire, Sleep questionnaire, Depression questionnaire, Quality of life and financial questionnaire
  Alpha Stim AID cranial electrotherapy stimulation: - 60 minutes of cranial electrotherapy stimulation via Alpha Stim AID once per day, for a minimum of 6 and maximum of 12 weeks.
  Pregnancy test: - Pregnancy test (day 1)
  Anxiety questionnaire: - GAD-7 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life questionnaire: - EQ-5D-5L (day 1, week 4, week 6, week 8, week 12 and week 24)
  Work and social questionnaire: - WASA (day 1, week 4, week 6, week 8, week 12 and week 24)
  Sleep questionnaire: - Athens (day 1, week 4, week 6, week 8, week 12 and week 24)
  Depression questionnaire: - PHQ-9 (day 1, week 4, week 6, week 8, wee
Arm/Group | Cranial Electrotherapy Stimulation at 100 uA for 60 Minutes
Number analyzed (Participants) | 161
Participants | 102

2. Secondary Outcome: Cost Effectiveness in Generalised Anxiety Disorder Compared to Current Treatment Approaches
Description: The secondary objective of this study is to evaluate the cost effectiveness of treatment with Alpha-Stim AID Cranial Electrotherapy Stimulations (CES) for participants with a primary working diagnosis of generalised anxiety disorder (GAD), in terms of health and social care service cost, and patient cost, from baseline to week 24, following previous treatment with low intensity psychological therapy intervention. The health and social care service cost and patient cost will be aggregated to determine the QALY (quality adjusted life year) value of the intervention. QALYs are used by the National Institute for Clinical Excellence (NICE) in the United Kingdom to determine the cost effectiveness of a treatment, and to determine whether it should be made available free at point of use in the National Health Service (NHS).
Time Frame: 24 weeks
Population: Cost savings per patient of treatment with Alpha-Stim versus treatment as usual
Measure: Number (95% Confidence Interval); unit: Pound sterling
Groups:
- Cranial Electrotherapy Stimulation at 100 uA for 60 Minutes: Alpha Stim AID cranial electrotherapy stimulation, Pregnancy test, Anxiety questionnaire, Quality of life questionnaire, Work and social questionnaire, Sleep questionnaire, Depression questionnaire, Quality of life and financial questionnaire
  Alpha Stim AID cranial electrotherapy stimulation: - 60 minutes of cranial electrotherapy stimulation via Alpha Stim AID once per day, for 6 to 12 weeks.
  Pregnancy test: - Pregnancy test (day 1)
  Anxiety questionnaire: - GAD-7 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life questionnaire: - EQ-5D-5L (day 1, week 4, week 6, week 8, week 12 and week 24)
  Work and social questionnaire: - WASA (day 1, week 4, week 6, week 8, week 12 and week 24)
  Sleep questionnaire: - Athens (day 1, week 4, week 6, week 8, week 12 and week 24)
  Depression questionnaire: - PHQ-9 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life and financial questionnaire: - CSRI (day 1, week 12 and week 24)
Arm/Group | Cranial Electrotherapy Stimulation at 100 uA for 60 Minutes
Number analyzed (Participants) | 161
Pound sterling | 540 [327 to 648]

3. Secondary Outcome: Clinical Effectiveness in Depression as Measured by Reduction of at Least 6 Points in Scores on the Personal Health Questionnaire (PHQ-9)
Description: The third objective of this study is to evaluate the clinical effectiveness of treatment with Alpha-Stim AID Cranial Electrotherapy Stimulations (CES) for depression in participants with a primary working diagnosis of generalised anxiety disorder (GAD), in terms of reliable improvement (a 6 point reduction in scores on the PHQ-9) or recovery (a score of 9 or less and at least a 6 point drop on the PHQ-9), from baseline to week 24, following previous treatment with low intensity psychological therapy intervention.
Time Frame: 24 weeks
Population: Number of participants with at least reliable improvement in depression symptoms
Measure: Count of Participants; unit: Participants
Arm/Group | Cranial Electrotherapy Stimulation at 100 uA for 60 Minutes
Number analyzed (Participants) | 161
Participants | 80

4. Secondary Outcome: Clinical Effectiveness in Insomnia as Measured by at Least a 50% Reduction in Score on the Athens Insomnia Scale (AIS)
Description: The fourth objective of the tertiary objective of this study is to evaluate the clinical effectiveness of treatment with Alpha-Stim AID Cranial Electrotherapy Stimulations (CES) for insomnia in participants with a primary working diagnosis of generalised anxiety disorder (GAD), in terms of reliable improvement (at least a 50% reduction in scores on the AIS), and recovery (a score of less than 4 and a reduction of at least 50% in AIS score), from baseline to week 24, following previous treatment with low intensity psychological therapy intervention.
Time Frame: 24 weeks
Population: Number of participants experiencing at least reliable improvement in sleep
Measure: Count of Participants; unit: Participants
Groups:
- Cranial Electrotherapy Stimulation at 100 uA for 60 Minutes: Alpha Stim AID cranial electrotherapy stimulation, Pregnancy test, Anxiety questionnaire, Quality of life questionnaire, Work and social questionnaire, Sleep questionnaire, Depression questionnaire, Quality of life and financial questionnaire
  Alpha Stim AID cranial electrotherapy stimulation: - 60 minutes of cranial electrotherapy stimulation via Alpha Stim AID once per day, for 6 to 12 weeks.
  Pregnancy test: - Pregnancy test (day 1)
  Anxiety questionnaire: - GAD-7 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life questionnaire: - EQ-5D-5L (day 1, week 4, week 6, week 8, week 12 and week 24)
  Work and social questionnaire: - WASA (day 1, week 4, week 6, week 8, week 12 and week 24)
  Sleep questionnaire: - Athens(day 1, week 4, week 6, week 8, week 12 and week 24)
  Depression questionnaire: - PHQ-9 (day 1, week 4, week 6, week 8, week 12 and week 24)
  Quality of life and financial questionnaire: - CSRI (day 1, week 12 and week 24)
Arm/Group | Cranial Electrotherapy Stimulation at 100 uA for 60 Minutes
Number analyzed (Participants) | 161
Participants | 48

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Cranial Electrotherapy Stimulation
All-Cause Mortality (participants affected / at risk) | 0/161
Serious Adverse Events (participants affected / at risk) | 0/161
Other Adverse Events (participants affected / at risk) | 4/161
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cranial Electrotherapy Stimulation (N=161)
Headache and insomnia (Product Issues) | 2 (2) — Headache and insomnia are known possibilities of CES if the current is set too high for the participant to used too close to bedtime.
Nausea (Gastrointestinal disorders) | 1 (1) — Nausea is a known possibility of CES treatment if the current is set too high for the participants
Strange feeling after use (General disorders) | 1 (1) — Participant was nonspecific regarding the event.

LIMITATIONS AND CAVEATS:
Sample was not an RCT and did not have a placebo control group. Lack of ethnic diversity in the sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT02901080/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT02901080/ICF_001.pdf